CLINICAL TRIAL: NCT02870205
Title: A Double-Blind, Randomized, Parallel-Group Seasonal Allergic Rhinitis (SAR) Study to Evaluate the Efficacy, Safety and Tolerability of GSP 301 Nasal Spray Compared With Placebo Nasal Spray and Individual Monotherapy Formulations (Olopatadine Hydrochloride Nasal Spray and Mometasone Furoate Nasal Spray) in Adult and Adolescent Subjects (12 Years of Age and Older)
Brief Title: Efficacy and Safety of GSP 301 Nasal Spray in the Treatment of Seasonal Allergic Rhinitis (SAR)
Acronym: GSP 301-304
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glenmark Specialty S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GPL/CT/2015/004/III; Study Number: GSP 301-304 (Other: Glenmark Specialty S.A.)
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Results first posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Seasonal Allergic Rhinitis (SAR)
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- GSP 301 NS (Experimental)
  Interventions: Drug: GSP 301 NS
- GOM-NS (Active Comparator)
  Interventions: Drug: GOM-NS
- GMM-2 NS (Active Comparator)
  Interventions: Drug: GMM-2 NS
- GSP 301 placebo NS (Placebo Comparator)
  Interventions: Drug: GSP 301 placebo NS

INTERVENTIONS:
Drug: GSP 301 NS — 2 spray in each nostril twice daily for 14 days
  Arms: GSP 301 NS
Drug: GOM-NS — 2 spray in each nostril twice daily for 14 days
  Arms: GOM-NS
Drug: GMM-2 NS — 2 spray in each nostril twice daily for 14 days
  Arms: GMM-2 NS
Drug: GSP 301 placebo NS — 2 spray in each nostril twice daily for 14 days
  Arms: GSP 301 placebo NS

SUMMARY:
Study to evaluate the efficacy, safety and tolerability of GSP 301 NS compared with placebo NS and individual monotherapy formulations for the treatment of Seasonal Allergic Rhinitis (subjects 12 years of age and older)

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females who are 12 years of age and older.
* Documented clinical history of SAR (for at least 2 years preceding the Screening Visit [Visit 1]) with exacerbations (clinical evidence of active symptoms) for the relevant seasonal allergen during the Fall or mountain cedar allergy seasons (e.g., ragweed or mountain cedar pollen)
* A 12-hour rTNSS ≥8 out of a possible 12 and a congestion score ≥2 for the AM assessment at the Screening Visit (Visit 1).

Exclusion Criteria:

* Pregnant or lactating women.
* History of anaphylaxis and/or other severe local reaction(s) to skin testing.
* History of positive test for HIV, Hepatitis B or Hepatitis C infection.
* Documented evidence of acute or significant chronic sinusitis or chronic purulent postnasal drip.
* Subjects with an active pulmonary disorder or infection.
* Subjects with posterior subcapsular cataracts or glaucoma
* Plans to travel outside the known pollen area for the investigational site for 24 hours or longer during the last 7 days of the run-in period.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1176 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudeesh Tantry, PhD, Study Director — Glenmark Pharmaceuticals Ltd
Locations (43):
- United States (43):
  - Investigational Site 406, Mission Viejo, California
  - Investigational Site 414, Orange, California
  - Investigational Site 435, San Diego, California
  - Investigational Site 420, Centennial, Colorado
  - Investigational Site 444, Colorado Springs, Colorado
  - Investigational Site 428, Aventura, Florida
  - Investigational Site 412, Miami, Florida
  - Investigational Site 436, Bethesda, Maryland
  - Investigational Site 432, South Dartmouth, Massachusetts
  - Investigational Site 426, Minneapolis, Minnesota
  - Investigational Site 403, Plymouth, Minnesota
  - Investigational Site 443, Columbia, Missouri
  - Investigational Site 441, Rolla, Missouri
  - Investigational Site 440, St Louis, Missouri
  - Investigational Site 405, Bellevue, Nebraska
  - Investigational Site 434, Skillman, New Jersey
  - Investigational Site 408, Rochester, New York
  - Investigational Site 418, Rockville Centre, New York
  - Investigational Site 402, High Point, North Carolina
  - Investigational Site 427, Raleigh, North Carolina
  - Investigational Site 419, Cincinnati, Ohio
  - United States 404, Cincinnati, Ohio
  - United States 407, Edmond, Oklahoma
  - Investigational Site 410, Oklahoma City, Oklahoma
  - Investigational Site 424, Tulsa, Oklahoma
  - Investigational Site 411, Pittsburgh, Pennsylvania
  - Investigational Site 416, Spartanburg, South Carolina
  - Investigational Site 415, Austin, Texas
  - Investigational Site 442, Austin, Texas
  - Investigational Site 417, Boerne, Texas
  - Investigational Site 421, Dallas, Texas
  - Investigational Site 430, Dallas, Texas
  - Investigational Site 431, El Paso, Texas
  - Investigational Site 433, Kerrville, Texas
  - Investigational Site 422, New Braunfels, Texas
  - Investigational Site 401, San Antonio, Texas
  - Investigational Site 413, San Antonio, Texas
  - Investigational Site 425, San Antonio, Texas
  - Investigational Site 437, San Antonio, Texas
  - Investigational Site 400, Waco, Texas
  - Investigational Site 409, Waco, Texas
  - Investigational Site 423, Draper, Utah
  - Investigational Site 439, Greenfield, Wisconsin

REFERENCES:
- [Derived] Gross GN, Berman G, Amar NJ, Caracta CF, Tantry SK. Efficacy and safety of olopatadine-mometasone combination nasal spray for the treatment of seasonal allergic rhinitis. Ann Allergy Asthma Immunol. 2019 Jun;122(6):630-638.e3. doi: 10.1016/j.anai.2019.03.017. Epub 2019 Mar 22. PMID 30910440
- See also: Poster presentation at the "2017 Annual Scientific Meeting of the American College of Allergy, Asthma, and Immunology" — http://epostersonline.com/acaai2017/node/1113

RESULTS

PARTICIPANT FLOW:
Groups:
- GSP 301 Placebo NS; GSP 301 NS; Olopatadine HCl NS; Mometasone Furoate NS: 2 sprays/nostril twice daily for 14 days
Period: Overall Study
Arm/Group | GSP 301 Placebo NS | GSP 301 NS | Olopatadine HCl NS | Mometasone Furoate NS
Started | 294 | 294 | 294 | 294
Completed | 284 | 289 | 287 | 287
Not Completed | 10 | 5 | 7 | 7

BASELINE CHARACTERISTICS:
Population: GSP 301 placebo NS: Due to repeated participation of same subject in 2 seasons, only 1 participation (fall period) was included; Mometasone furoate NS: 1 subject received wrong kit and was excluded; GSP 301 NS and olopatadine HCl NS: Due to coinciding participation of same subject at 2 different sites, both participation's were excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | GSP 301 Placebo NS | GSP 301 NS | Olopatadine HCl NS | Mometasone Furoate NS | Total
Number analyzed (Participants) | 293 | 293 | 293 | 293 | 1172
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (14.93) | 39.9 (14.91) | 39.9 (14.62) | 39.2 (14.86) | 39.6 (14.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 202 | 189 | 170 | 737
  Male | 117 | 91 | 104 | 123 | 435

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average AM and PM Subject-reported 12-hour Reflective Total Nasal Symptom Score (rTNSS)
Description: The Reflective Total Nasal Symptom Score (rTNSS) was assessed by 12-hour reflective scoring of the severity of four nasal symptoms (rhinorrhea, sneezing, nasal congestion, nasal itching). Symptom scores ranged from 0 (no signs/symptoms evident) to 3 (severe signs/symptoms that is hard to tolerate). The rTNSS was calculated as the sum of the subject-reported severity scores for nasal symptoms, and value ranged from 0 (no signs/symptoms evident) to 12 (severe signs/symptoms that is hard to tolerate).
Time Frame: Baseline and day 14
Population: The FAS was defined as all subjects who were randomized and received at least one dose of investigational product and had at least one post-baseline primary efficacy assessment. This was the primary analysis set for efficacy analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GSP 301 Placebo NS | GSP 301 NS | Olopatadine HCl NS | Mometasone Furoate NS
Number analyzed (Participants) | 293 | 292 | 293 | 294
units on a scale
  Baseline | 10.3 (1.2) | 10.1 (1.2) | 10.2 (1.3) | 10.2 (1.3)
  Change from baseline to end of treatment | -2.9 (3.2) | -4.3 (3.1) | -3.6 (3.3) | -3.5 (3.5)
Statistical Analysis 1: Comparison: GSP 301 Placebo NS vs GSP 301 NS; Test type: Superiority; p < 0.001, ANCOVA — GSP 301 NS vs GSP 301 placebo NS comparison for rTNSS was tested at 0.05 significance level
Statistical Analysis 2: Comparison: GSP 301 NS vs Olopatadine HCl NS; Test type: Superiority; p = 0.028, ANCOVA
Statistical Analysis 3: Comparison: GSP 301 NS vs Mometasone Furoate NS; Test type: Superiority; p = 0.019, ANCOVA
Statistical Analysis 4: Comparison: GSP 301 Placebo NS vs Olopatadine HCl NS; Test type: Superiority; p < 0.001, ANCOVA
Statistical Analysis 5: Comparison: GSP 301 Placebo NS vs Mometasone Furoate NS; Test type: Superiority; p = 0.002, ANCOVA

ADVERSE EVENTS:
Time Frame: The AEs and SAEs were collected from the time of signing the informed consent form until the end of study i.e., 7-10 days of screening and placebo run-in and 14 days of treatment.
Description: Mometasone furoate NS: 1 subject received wrong kit and was excluded
Arm/Group | GSP 301 Placebo NS | GSP 301 NS | Olopatadine HCl NS | Mometasone Furoate NS
Serious Adverse Events (participants affected / at risk) | 1/294 | 0/294 | 2/294 | 1/293
Other Adverse Events (participants affected / at risk) | 0/294 | 0/294 | 0/294 | 0/293
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSP 301 Placebo NS (N=294) | GSP 301 NS (N=294) | Olopatadine HCl NS (N=294) | Mometasone Furoate NS (N=293)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per the agreement, Sponsor reserves the right for publishing trial results and the Investigator cannot publish without written consent from the CRO/Sponsor.